CLINICAL TRIAL: NCT02607267
Title: The Importance of the Edmonton Obesity Score System in Predicting Postoperative Outcome and 30 Day Mortality After Metabolic Surgery
Brief Title: Edmonton Obesity Staging System: Post-operative Outcome and 30-day Mortality
Status: Completed | Type: Observational
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, MD, Sana Klinikum Offenbach
Other Study IDs: FF 83/2015
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Complications; Other Complications of Other Bariatric Procedure
Keywords: EOSS; Metabolic Surgery; postoperative outcome; 30 - day mortality
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laparoscopic Roux en Y Gastric Bypass: patients undergoing LRYGB, being the first surgical treatment for severe obesity
  Interventions: Other: LSG and LRYGB
- laparoscopic Sleeve Gastrectomy: patients undergoing LSG, being the first surgical treatment for severe obesity
  Interventions: Other: LSG and LRYGB

INTERVENTIONS:
Other: LSG and LRYGB — The role of the Edmonton Obesity Staging System in predicting post-operative outcome and 30-day mortality after metabolic surgery (LSG and LRYGB)

SUMMARY:
The Edmonton Obesity Staging System (EOSS) is a more comprehensive measure of obesity-related diseases and predictor of mortality than BMI or waist circumference. The aim of this study is to determine whether the EOSS is also important in predicting post - operative outcome and 30-day mortality after metabolic surgery.

DETAILED DESCRIPTION:
From October 2014 to December 2015 the investigators conducted a prospective data collection on patients undergoing either laparoscopic sleeve gastrectomy (LSG) or laparoscopic Gastric Bypass (Laparoscopic Roux-en-Y-Gastric Bypass (LRYGB) and Omega-Loop-Gastric-Bypass (LOLGB)), being the first surgical treatment for severe obesity. Preoperative EOSS by Sharma et al. was applied to all patients by two different evaluators. Data collection included the following: gender, age, body mass index, waist circumference, waist to hip ratio, comorbidities, early - postoperative complications, readmission rates and 30 - day mortality. Follow-up was performed in all patients up to 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing either LSG or LRYGB, being the first surgical treatment for severe obesity

Exclusion Criteria:

* bariatric surgery in the anamnesis

Ages: 19 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing either LSG, LRYGB or LOLGB, being the first surgical treatment for severe obesity
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
postoperative outcome related to EOSS | 30 days after surgery

SECONDARY OUTCOMES:
postoperative complications related to EOSS | 30 days after surgery
readmission rates related to EOSS | 30 days after surgery
age related to postoperative complications | 30 days after surgery
BMI related to postoperative complications | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stier, MD, Study Director — Sana Klinikum Offenbach
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Hesse, Germany

REFERENCES:
- [Background] Kuk JL, Ardern CI, Church TS, Sharma AM, Padwal R, Sui X, Blair SN. Edmonton Obesity Staging System: association with weight history and mortality risk. Appl Physiol Nutr Metab. 2011 Aug;36(4):570-6. doi: 10.1139/h11-058. Epub 2011 Aug 14. PMID 21838602
- [Background] Padwal RS, Pajewski NM, Allison DB, Sharma AM. Using the Edmonton obesity staging system to predict mortality in a population-representative cohort of people with overweight and obesity. CMAJ. 2011 Oct 4;183(14):E1059-66. doi: 10.1503/cmaj.110387. Epub 2011 Aug 15. PMID 21844111
- [Background] Gill RS, Karmali S, Sharma AM. The potential role of the Edmonton obesity staging system in determining indications for bariatric surgery. Obes Surg. 2011 Dec;21(12):1947-9. doi: 10.1007/s11695-011-0533-8. No abstract available. PMID 22002510
- [Result] Sharma AM, Kushner RF. A proposed clinical staging system for obesity. Int J Obes (Lond). 2009 Mar;33(3):289-95. doi: 10.1038/ijo.2009.2. Epub 2009 Feb 3. PMID 19188927